CLINICAL TRIAL: NCT05440747
Title: A Multicenter, Observational Register Study of Treatment Free Remission in Patients With Chronic Myeloid Leukemia (CML-CP)
Brief Title: Treatment Free Remission (TFR) in CML Patients （CML-CP）Study
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, WENG Jian yu, Professor, Guangdong Provincial People's Hospital
Other Study IDs: GDPH-CML-TFR-2020-12
Record Dates: First submitted 2022-04-02; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia; Treatment-free Remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly diagnosed CML-CP patients: Treat with TKI (Imatinib or Flumatinib or Nilotinb or Dasatinib).
  Interventions: Other: TFR(Treatment-Free Remission)
- Patients with suboptimal response: 1. Treat with original TKI
  2. Treat with original TKI combined with interferon/thymosin;
  3. Replace other TKI ;
  4. Replace other TKI and combined with interferon/thymosin.
  Interventions: Other: TFR(Treatment-Free Remission)

INTERVENTIONS:
Other: TFR(Treatment-Free Remission) — Withdrawal TKIs(Tyrosine kinase inhibitors: Imatinib or Flumatinib or Nilotinb or Dasatinib)

SUMMARY:
Improving the quality of life and achieving Treatment-Free Remission(TFR) is a long-term goal of treatment in CML-CP patients, and deep molecular response (DMR) is necessary to achieve TFR. Cording to the historical literature, it is reported that patients with CML-CP take MMR as the therapeutic target, and the acquisition rate of DMR under long-term TKI treatment is 50%. The 2-year success rate of TFR patients was 50%. Therefore, maybe only 25% of patients with CML can successfully stop the drug for a long time. It cannot meet the withdrawal needs of patients with long-term drug survival.

This study is to design a real-world observational registration study for optimal effect. On the premise of taking DMR as the target decision, through initial treatment intervention, improve the DMR rate, which will promote clinical practice, so as to improve the 2-year TFR rate of cml-cp patients. This study is a multicenter, observational, prospective registry to identify the optimal treatment for achieving TFR in CML patients. In this study, the investigators will assess the deep molecular response after 12 months of treatment and the 2-year treatment-free remission rate (TFR 2y) after drug discontinuation.

Eligible participants with CML-CP can be enrolled. The observation period of all participants is at least 60 months, of which the first 36 months is the shortest treatment period, and the last 24 months is the TFR observation period after TKIs (Imatinib/Flumatinib/Nilotinb/ Dasatinib) withdrawal. During the treatment phase, participants can receive TKIs ± IFN (or other treatments) as first-line/second-line treatment, and the treatment plan will be adjusted according to the molecular response. Patients should accept TKI treatment for at least 3 years or more, and MR4/MR4.5 should achieve at least 2 years before discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged >=14 years old male and female;
* 2) Patients with Ph+ CML-CP should meet any of the following conditions;

  1. Newly diagnosed Patients with CML-CP;
  2. The CML-CP patients who treated with TKI (Imatinib, Nilotinib, Dasatinib and Flumatinib) are not achieved optimal （BCR-ABLIS>10% in 3 months, BCR-ABLIS>1% in 6 months, BCR-ABLIS>0.1% in 12 months or BCR-ABLIS>0.01% in 24 months ）or intolerance to these TKIs; The definition of the confirmed diagnosis: Bone marrow cytogenetics Ph chromosome t(9;22) positive and/or BCR-ABL fusion gene positive by FISH, and/or BCR-ABL fusion gene positive(>10%) by Q-PCR ;
* 3) Never received stem cell transplantation before enrollment;
* 4) Female patients with fertility have a negative pregnancy test (within 7 days before enrollment).

All Patients with TFR requeirement should provid written informed consent before enrollment.

Exclusion Criteria:

1. T315I mutation is known;
2. Received stem cell transplantation before enrollment;
3. With other malignant tumors and need active intervention;
4. Those who are unable to follow the protocol steps or follow up on time;
5. Eastern Cooperative Oncology Group physical performance score (ECOG PS) >=3;
6. Other situations deemed unsuitable by the researcher.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants should older than 14 years old, and Newly diagnosed with CML-CP or had been treated with TKI (Imatinib, Nilotinib, Dasatinib and Flumatinib) are not achieved optimal (BCR-ABLIS>10% in 3 months, BCR-ABLIS>1% in 6 months, BCR-ABLIS>0.1% in 12 months or BCR-ABLIS>0.01% in 24 months) or intolerance to these TKIs.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Deep molecular response(DMR) rate of 12 months | The 12th month
  DMR is defined by IS BCR-ABL/ABL achieve MR4.0(≤0.01%)
Treatment-Free Remission(TFR) rate of 2 years | The second year
  The proportion of drug withdrawal

SECONDARY OUTCOMES:
TFR rate | The 6months、12months
  TFR rate of 6/12months，Median duration of TFR
DMR rate | The 24/36/48/60 months
  DMR rate of 24/36/48/60 months, Median duration of DMR, DMR is defined by IS BCR-ABL/ABL achieve MR4.0
DMR persistence rate in 2 years | 2 years
  DMR is defined by IS BCR-ABL/ABL achieve MR4.0
Disease progression rate , time to progression | The whole study, up to 7 years
  Time and proportion from diagnosis to disease progression to AP or BC
Loss of Major Molecular Remission(MMR-loss IS BCR-ABL≥0.1%） | TFR phase in the study, up to 2 years
  Time and proportion from discontinuation to loss of MMR in TFR phase up to 2 years.
Re-Major Molecular Remission | The TFR phase, up to 2 years
  Time and proportion from restarting therapy after MMR-lose to obtain MMR through TFR phase.
Treatment-related safety | The whole study , up to 7 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Patient Report Outcome（PRO） | Every 3 months in the whole enrollment period, up to 7 years
  EORTCQLQ-CML-24 survey every 3 months in the whole enrollment period

OTHER OUTCOMES:
Clonal evolution in CML patients without optimal efficacy | After participants loss optimal efficacy in milestone,and once a years after that, up to 7 years
  Bone marrow karyotype analysis once a year in the patients without optimal efficacy in milestone through study completion
Resistant mutation rate | The whole study, up to 7 years
  Molecular Mutation Examination（qPCR) once a year in patient without optimal efficacy through study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Jianyu, PhD, Study Chair — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: Yes
After the study was complete, IPD will be uploaded as an supplementary data of the research paper. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
Supporting Information: CSR